CLINICAL TRIAL: NCT02663193
Title: A Multicenter, Two-arm, Prospective, Observational Study to Characterize the Tolerability of Treatment With Enzalutamide or Abiraterone Acetate (With Prednisone) for Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: Real-World Study of Enzalutamide and Abiraterone Acetate (With Prednisone) Tolerability
Acronym: REAAcT
Status: Completed | Type: Observational
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108103; 212082PCR4038 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Observational study; Enzalutamide; Abiraterone Acetate; Prednisone; Tolerability
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Enzalutamide Group: Participants who are receiving enzalutamide in a clinical practice setting will be observed for tolerability and quality of life.
  Interventions: Other: No Intervention
- Abiraterone Acetate plus Prednisone group: Participants who are receiving abiraterone acetate in combination with prednisone in a clinical practice setting will be observed for tolerability and quality of life.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Participants who are receiving enzalutamide or abiraterone acetate in combination with prednisone in a clinical practice setting will be observed for tolerability and quality of life.

SUMMARY:
The purpose of this study is to characterize the tolerability profiles of enzalutamide and abiraterone acetate (with prednisone) -with specific focus on central nervous system (CNS) tolerability-and quality of life (QoL) after approximately 2 months of participants starting treatment with one of these agents for metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This is a multicenter (more than one study site), open-label (all people know the identity of the intervention), prospective, observational study to characterize the tolerability profile of treatment and quality of life (QoL) in participants receiving enzalutamide or abiraterone acetate (with prednisone) in a clinical practice setting. Approximately 100 male participants will be enrolled into this study, 50 participants will be recruited to each treatment arm. Participants will complete 2 scheduled on-site visits (Baseline and Month 2). Participants will primarily be observed for tolerability profiles of enzalutamide and abiraterone acetate (with prednisone) and safety over an observational period of 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Male 18 years of age or older
* Have confirmed metastatic adenocarcinoma of the prostate
* Are starting treatment with enzalutamide or abiraterone acetate (with prednisone) for metastatic castration-resistant prostate cancer (mCRPC) at the full recommended dose per each drug's respective prescribing information (PI)
* Have an Eastern Cooperative Oncology Group Performance Status score of 0 or 1
* Sign written informed consent

Exclusion Criteria:

* Have a pre-existing central nervous system (CNS) condition (including, but not limited to, history of stroke or dementia) that, in the participating physician's judgment, would preclude participation in the study
* Have known mental illness including, but not limited to, major depressive disorder, general anxiety disorder, or bipolar disorder that, in the participating physician's opinion, could significantly confound the patient-reported outcome (PRO) assessments
* Have a history of or ongoing seizure disorder
* Have severe hepatic impairment (Child-Pugh Class C)
* Have an active infection (example, human immunodeficiency virus [HIV], viral hepatitis) or other medical condition that would contraindicate the use of prednisone/prednisolone (systemic glucocorticoid)
* Have known alcohol or other substance abuse disorder
* Are routinely taking medication-including, but not limited to, over-the-counter medications, supplements, medical marijuana or prescription pain medication-that is known to cause mental confusion or sedation or are using any of the medications
* Are routinely taking systemic glucocorticoids (example, prednisone, prednisolone, dexamethasone) at a dosage higher than the equivalent of prednisone 10 milligram (mg) daily
* Are currently using or have previously used chemotherapy for any cancer including mCRPC
* Are concurrently using any first-generation androgen-receptor blocker (example, bicalutamide, flutamide, nilutamide) for mCRPC
* Have previously taken enzalutamide or abiraterone acetate with prednisone
* Are not capable of completing tests using a computerized system or completing a participant survey

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have a confirmed metastatic adenocarcinoma of the prostate will receive either enzalutamide or abiraterone acetate with prednisone for the treatment at the discretion of their treatment physician and in accordance with clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2015-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Cogstate Tests at Month 2 | Baseline and Month 2
  The Cogstate computerized cognitive test battery will be used as the assessment tool in this study. Overall, Cogstate measures a range of cognitive functions (example, psychomotor and memory function) using a number of different tests (example, choice reaction time, one-back memory). This battery of tests was chosen because it has been shown to be sensitive to very small cognitive changes and has been tested in cancer participants after chemotherapy.
Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 at Month 2 | Baseline and Month 2
  The EORTC QLQ-C30 is a questionnaire developed to assess the quality of Life (QoL) of cancer participants. The QLQ-C30 incorporates 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social); 3 symptom scales (fatigue, pain, and nausea and vomiting); and a global health and QoL scale.
Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue subscale (FACIT-Fatigue) at Month 2 | Baseline and Month 2
  The FACIT Measurement System is a collection of health-related QoL questionnaires targeted to the management of chronic illness. The fatigue subscale (FACIT-Fatigue) is a validated, 13-item questionnaire that assesses fatigue in people being treated for a chronic illness.
Change From Baseline in Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) at Month 2 | Baseline and Month 2
  The FACT-Cog is a validated, 37-item, subjective neuropsychological instrument designed to evaluate cancer participants perceived cognitive deterioration on their quality of life.
Participant or Caregiver Observational Questionnaire (Survey) | Baseline
  If a participant has a regular caregiver, the participating physician will ask the caregiver to complete an optional observational, sponsor-developed questionnaire (survey) pertaining to his/her perception of the participants tolerability of treatment and QoL.
Participant or Caregiver Observational Questionnaire (Survey) | Month 2
  If a participant has a regular caregiver, the participating physician will ask the caregiver to complete an optional observational, sponsor-developed questionnaire (survey) pertaining to his/her perception of the participants tolerability of treatment and QoL.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up (Approximately 2 Months)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (20):
- United States (20):
  - Homewood, Alabama
  - La Mesa, California
  - Wheat Ridge, Colorado
  - Daytona Beach, Florida
  - Indianapolis, Indiana
  - Jeffersonville, Indiana
  - Saint Clair Shores, Michigan
  - Englewood, New Jersey
  - Lawrenceville, New Jersey
  - Morristown, New Jersey
  - Poughkeepsie, New York
  - Syracuse, New York
  - Middleburg Heights, Ohio
  - Springfield, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Lancaster, Pennsylvania
  - Charleston, South Carolina
  - Myrtle Beach, South Carolina
  - San Antonio, Texas
  - Virginia Beach, Virginia